CLINICAL TRIAL: NCT01981733
Title: A Study to Determine the Effects of a Novel Method for Improving Lower Limb Blood Flow in Healthy Adult Volunteers
Brief Title: Improving Lower Limb Blood Flow in Healthy Adult Volunteers
Acronym: THRIVE-1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Basic Science
Other Study IDs: THRIVE-1
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental)
  Interventions: Device: geko

INTERVENTIONS:
Device: geko — The geko is a neuromuscular stimulator device, which when applied stimulates the common peroneal nerve
  Other Names: geko TM

SUMMARY:
The THRIVE-1 study will examine novel methods for enhancing blood flow in the lower limb using electrical stimulation. Increases in lower limb blood flow improve venous return and thereby reduce venous stasis. Since stasis is one of the compounding factors in the development of deep vein thrombosis, the risk of developing thrombosis should theoretically be proportionally reduced. This technique may prove to be a useful tool in preventing and reducing the incidence of deep vein thrombosis in both medical and surgical patients together with passengers undertaking significant duration travel (as travel - related deep vein thrombosis is not exclusively related to flying).

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general health and fitness.
2. Aged between 18 and 65 years.
3. Free of significant abnormal findings as determined by medical history (specifically an absence of DVT or haematological disorders or indications), screening physical examination, vital signs (sitting blood pressure, sitting pulse rate, sitting respiratory rate and body temperature) and duplex ultrasound within 48 hours prior to commencement of the each study phase.
4. BMI between 18 and 34
5. No history or signs of drug abuse (including alcohol), licit or illicit.
6. Has not to used any medications (prescribed or over-the-counter including herbal remedies) judged to be significant by the Principal Investigator during the thirty (30) days preceding the study, and agrees not to use any medications during the course of the study without informing the Research Team.
7. Able to understand the Volunteer Information Sheet and signed the written Informed Consent Forms.
8. Able and willing to follow the Protocol requirements.

Exclusion Criteria:

1. Any evidence of organ dysfunction, or any clinically significant deviation from normal in the physical determinations.
2. History or signs of haematological disorders (especially in relation to clotting or coagulation or previous Deep or superficial vein thrombosis/pulmonary embolism).
3. Peripheral arterial disease (ABPI < 0.9), varicose veins or lower limb ulceration.
4. Musculoskeletal disorders (such as pain during exercise of lower limb).
5. Recent surgery (such as abdominal, gynaecological, hip knee replacement).
6. Recent trauma to lower limb.
7. Chronic Obesity (BMI Index >34).
8. Pregnancy.
9. Any Medication judged to be significant by the Principal Investigator (such as anticoagulants, agents with significant vasoactive activity, Oestrogen pill, 'morning-after pill' or HRT).
10. Tobacco consumption
11. History of disorders of the gastrointestinal, hepatic, renal, cardiovascular, endocrine, neurological, dermatological, rheumatologic, metabolic (including diabetes), psychiatric, haematological (especially in relation to clotting or coagulation), or systemic disease judged to be significant.
12. A pulse rate of less than 50 beats/minute, a sitting systolic blood pressure >160 or <80 mmHg and/or a sitting diastolic pressure of >90 or <60 mmHg.
13. Any significant illness during the four (4) weeks preceding the screening period of the study.
14. Any contraindication to blood sampling.
15. Donation of blood during the eight (8) weeks preceding the screening period of the study or during the investigation.
16. Participation in any clinical study during the 8 weeks preceding the dosing period of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in blood flow and volume, together with microcirculatory velocity were measured | 30 mins with 10 min washouts
  Changes in blood flow and volume, together with microcirculatory velocity were measured using laser Doppler flowmetry (Laser Doppler Perfusion & Temperature Monitor DRT4; Moor Instruments Ltd, UK) and colour flow duplex ultrasound (Philips IU22; Philips Healthcare, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Tucker, BSc PhD, Principal Investigator — St. Bartholomew's Hospital
Locations (1):
- St. Bartholomew's Hospital, London, United Kingdom